CLINICAL TRIAL: NCT01055717
Title: Bioavailability of Avenanthramide-Enriched Oats in Healthy Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: Agriculture and Agri-Food Canada (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB9306
Record Dates: First submitted 2010-01-25; First posted 2010-01-26 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2013-05

CONDITIONS: Healthy
Keywords: avenanthramide; enriched; oat; phytochemical; bioavailability
MeSH Terms: conditions — Gyrate Atrophy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo muffin made with no oats (Placebo Comparator)
  Interventions: Other: Avenanthramide-enriched oats
- Test muffin made with AV-enriched oats (Active Comparator)
  Interventions: Other: Avenanthramide-enriched oats

INTERVENTIONS:
Other: Avenanthramide-enriched oats — Single dose, 24 hour pharmacokinetic trial

SUMMARY:
This is a placebo-controlled, crossover study investigating the pharmacokinetic bioavailability of avenanthramides from avenanthramide-enriched oats and their in vivo metabolites in a cohort of healthy, older adults.

ELIGIBILITY:
Inclusion Criteria:

* Men and postmenopausal women
* BMI 18.5-29.9 kg/m2

Exclusion Criteria:

* Cigarette smoking and/or nicotine replacement use
* Use of cholesterol-lowering medications
* Use of blood pressure-lowering medications
* Use of any stomach acid-lowering medications
* Cardiovascular (heart) disease
* Gastrointestinal disease
* Kidney disease
* Endocrine disease: including diabetes, untreated thyroid disease
* Rheumatoid arthritis
* Active treatment for any type of cancer, except basal cell carcinoma, within 1 year prior to study admission
* Systolic blood pressure > 150 mm Hg and/or diastolic blood pressure > 95 mm Hg
* Regular use of oral steroids
* Regular daily intake of 2 or more alcoholic drinks
* Illicit drug use
* No fish oil supplements (including cod liver oil) for one month prior to study admission
* No dietary supplements, including those containing any vitamins, minerals, herbs, plant concentrates (including garlic, gingko, St. John's wort) or homeopathic remedies, for one month prior to study admission

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-03; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Levels of avenanthramides and their in vivo metabolites in blood, urine, and feces following the consumption of avenanthramide-enriched oats delivered in a baked muffin | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey B Blumberg, PhD, Principal Investigator — Jean Mayer USDA Human Nutrition Research Center on Aging at Tufts Unversity
Locations (1):
- Jean Mayer USDA Human Nutrition Research Center on Aging at Tufts University, Boston, Massachusetts, United States